CLINICAL TRIAL: NCT04971811
Title: Self-served Snack Study for Preschool Children
Brief Title: Effects of Energy Density on Self-served Snacks in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ChildFood601
Record Dates: First submitted 2021-07-20; First posted 2021-07-22 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Snacks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower-energy-dense Snack (Experimental): Test snack with lower-energy-dense snack food
  Interventions: Other: Snack with energy density less than 1.5 kcal/g
- Higher-energy-dense Snack (Experimental): Test snack with higher-energy-dense snack food
  Interventions: Other: Snack with energy density greater than 1.5 kcal/g

INTERVENTIONS:
Other: Snack with energy density less than 1.5 kcal/g — Snack meal with snack food having energy density less than 1.5 kcal/g
  Arms: Lower-energy-dense Snack
Other: Snack with energy density greater than 1.5 kcal/g — Snack meal with snack food having energy density greater than 1.5 kcal/g
  Arms: Higher-energy-dense Snack

SUMMARY:
The purpose of the study is to determine whether the energy density of snack foods affects the amounts that preschool children serve themselves and then consume. We will serve snacks that vary in energy density to preschool children in their childcare centers and measure the amount they serve themselves and consume. The results will have implications for guidance about the provision of snacks for preschool children and may help in identifying strategies for the prevention of obesity in children.

ELIGIBILITY:
Inclusion Criteria:

* Children who are enrolled in a scheduled classroom of the participating childcare centers
* Children who are between the ages of 4 and 6 years old at the time of enrollment

Exclusion Criteria:

* Children who have tested positive or are showing symptoms of COVID-19, or have recently had potential exposure with a person with COVID-19
* Children who are allergic to any of the foods served
* Children whose diets exclude any of the foods served
* Children who are absent from the childcare center on the acclimation day or both study days
* Children who are not able to serve themselves the two foods that are provided during the acclimation day

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Difference between interventions in the weight of self-served snack food | Study weeks 1 and 2
  Weight served of snack food in grams
Difference between interventions in the weight of snack food consumed | Study weeks 1 and 2
  Weight consumed of snack food in grams

SECONDARY OUTCOMES:
Difference between interventions in the volume of self-served snack food | Study weeks 1 and 2
  Volume served of snack food in milliliters (ml)
Difference between interventions in the volume of snack food consumed | Study weeks 1 and 2
  Volume consumed of snack food in milliliters (ml)
Difference between interventions in the energy of self-served snack food | Study weeks 1 and 2
  Energy served of snack food in kilocalories (kcal)
Difference between interventions in the energy of snack food consumed | Study weeks 1 and 2
  Energy consumed of snack food in kilocalories (kcal)

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No